CLINICAL TRIAL: NCT05104242
Title: A Feasibility Study Exploring the Impact of a Low Advanced Glycation End-product (AGE) Diet on Skin Autofluorescence (SAF) Levels in Kidney Transplant Recipients
Brief Title: Kidney Transplant Low-AGE Diet Study
Acronym: Transplant LAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: British Renal Society (Other); Kidney Care UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UHDB/2020/018
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Renal Transplant
MeSH Terms: interventions — Glycation End Products, Advanced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard diet - Control group (No Intervention): The standard diet will include energy intake of 30-35 kcal/kg of ideal body weight (IBW)/day and protein intake of 0.75 g/kg of IBW/day for females and 0.84 g/kg of IBW/day for males
- Low AGE diet - Intervention group (Experimental): The low AGE diet will be the same as the standard diet in terms of calories (i.e. 30-35 kcal/kg/day) and protein (0.75-0.84 g/kg/day). However, it will reduce the dietary AGE content by changing cooking methods in food preparation to avoid exposure to dry heat such as frying, broiling, grilling and roasting, and to favour cooking with lower temperatures and high-water content as in stewing, steaming, boiling and poaching. In addition, the low-AGE group will be instructed to choose foods with low content of AGEs based on a food choice list that will contain examples of foods commonly available in the UK to be chosen as "allowed," "moderate intake," or "occasional." The goal will be to reduce dietary AGE intake to less than 8000 kU/day.
  Interventions: Other: Diet low in Advanced Glycation End-Products (AGE)

INTERVENTIONS:
Other: Diet low in Advanced Glycation End-Products (AGE) — The low AGE diet will primarily consist in reducing the amount of AGEs in foods by changing cooking methods. Participants will also be advice to choose foods low in AGEs; however, the advice will be tailored to participants' food preferences
  Arms: Low AGE diet - Intervention group

SUMMARY:
The purpose of the present study is to test the feasibility of conducting a larger randomised controlled trial (RCT) which will investigate whether a diet low in toxins called advanced glycation end-products (AGEs) decreases skin autofluorescence (SAF; AGE accumulation in the skin) levels and improves heart and circulatory (i.e. cardiovascular) health in persons with a kidney transplant.

DETAILED DESCRIPTION:
Kidney transplantation is the optimal treatment option for end-stage kidney disease. Cardiovascular disease is the leading cause of death in persons with kidney disease, even after receiving a kidney transplant. Advanced glycation end-products (AGEs) are compounds that form naturally in our bodies from the chemical reaction of sugars with proteins. If the concentration of AGEs becomes excessive in our bloodstream, they can cause damage to almost every tissue and organ in our bodies, which eventually may lead to an increased risk of cardiovascular death and ill health. AGEs are also found naturally in foods and the content of AGEs in foods is increased considerably by using cooking methods that require high temperatures, such as frying, roasting and grilling.

Skin autofluorescence (SAF) is a relatively new, non-invasive, validated and easy to perform technique that measures the skin accumulation of AGEs. It has been reported that kidney transplant recipients have significantly lower SAF levels when compared to persons receiving dialysis; however, these are higher than the general population.

Because of the adverse outcomes (e.g. increased risk of death) strongly associated with higher levels of SAF, several options focused on reducing the accumulation of AGEs have been proposed. One of these promising interventions is the reduction of dietary intake of AGEs. It has been suggested that cooking techniques that avoid very high temperatures such as poaching, steaming, stewing and boiling can significantly reduce the AGE content of food when compared to frying, broiling, grilling and roasting. Several studies conducted in healthy overweight and/or obese volunteers, persons with diabetes and in those with chronic kidney disease and performing peritoneal dialysis have reported that reducing dietary AGE intake is associated with a reduction in blood levels of AGEs, suggesting that a low AGE diet may also be associated with a decrease in SAF. Nevertheless, most of the evidence regarding diet modifications to reduce dietary AGE intake is of low quality and therefore further studies are required. Furthermore, this simple dietary intervention has not been previously study in the kidney transplant population. Therefore, if this proposed feasibility study is successful, we will use these findings to identify ways to design future larger research projects to improve the care of persons with a kidney transplant.

This is a feasibility study that will be conducted in two parts:

Part 1:

This will be a randomised controlled trial (RCT) aiming to recruit 40 participants with a functional kidney transplant. Participants will be assigned to either a low AGE diet (intervention group) or a standard diet for persons with a kidney transplant (control group). Participants will be followed-up for 6 months and will receive precise oral and written advice on how to follow the diets. This advice will be tailored to their needs and food preferences.Adherence to both diets will be evaluated by means of a 3-day food diary (2 weekdays and 1 weekend day) every month.

The purpose of the control group is to show what would normally happen to AGE levels in the skin and compare it with what happens to AGE levels in the skin when persons with a kidney transplant follow a low AGE diet. Therefore, this will show if the low AGE diet is really responsible of the observations.

Potential participants will be approached by the Chief Investigator (a member of the transplant team), during routine follow-up appointments. After the participants have read and understand the Participant Information Sheet (PIS), and had sufficient time (at least 24 hours) to consider their participation in this study, we will ask them to sign a consent form, which shows their willingness to take part. We will then collect information from their medical records or direct interview about their age, ethnicity, medical conditions, educational level, employment and smoking status, medication, alcohol history, and information about their transplant and kidney disease.

During the first study assessment, we will:

* Measure the accumulation of toxins (AGEs) in the skin using a safe, quick (less than five minutes) and painless technique called skin autofluorescence. This involves placing the forearm on a piece of equipment that shines a light on the skin and measures the amount of light that is reflected back.
* Take routine blood samples and blood pressure.
* Ask participants to complete a quality of life questionnaire (EQ-5D-5L), a 3-day food diary (2 weekdays and 1 weekend day) to assess energy, fat and protein intake and a validated food frequency questionnaire to evaluate dietary AGE intake.
* Assess nutritional status using the validated 7-point scale Subjective Global Assessment.
* Measure weight, height, mid-arm circumference, triceps skinfold thickness, handgrip strength and aortic pulse wave velocity (a measure of cardiovascular health).

These same procedures and measurements will be conducted at 3 and 6 months of follow-up.

Part 2:

Once the RCT (Part 1) has finished, 10 participants from the intervention group and 5 from the control group (ensuring as far as possible that the sample includes a diverse representation of the study population), will be invited to take part in interviews asking questions about the acceptability and tolerability of the intervention (low AGE diet), as well as feedback about the study process.

Potential participants will be given or sent an invitation letter and PIS, have the study explained to them and consented separately. The interview will take place at a time and location convenient to the participants and will take about 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) with a functioning (not on dialysis) kidney transplant.
* More than 12 months post-transplant.
* Able and willing to give informed consent.
* Skin Autofluorescence levels above the general population mean value for age.

Exclusion Criteria:

* Persons with dark skin colour (i.e. Fitzpatrick skin colour type 5-6).
* Persons with malnutrition (Subjective Global Assessment [SGA] score <5).
* Pregnancy or breast feeding or intending pregnancy.
* Active infection.
* Active rejection.
* Persons with learning difficulties.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Johnson, Principal Investigator — University Hospitals of Derby and Burton NHS Foundation Trust
Locations (1):
- University Hospitals of Derby and Burton NHS Foundation Trust, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 48 kidney transplant recipients from the Department of Renal Medicine, Royal Derby Hospital were assessed for eligibility from February to April 2022.
Pre-assignment Details: Of the 48 kidney transplant recipients assessed for eligibility, 10 did not meet the inclusion criteria: 9 had skin autofluorescence levels below the general population mean value for age and 1 was classified as being malnourished according to the Subjective Global Assessment).
Groups:
- Standard Diet - Control Group: The control group was advised to follow their usual diet but aiming to achieve an energy intake of 25-35 kcal/kg/day, and a protein intake of 0.75 g/kg/day for females and 0.84 g/kg/day for males
- Low AGE Diet - Intervention Group: The intervention group was advised to follow a low-AGE diet which consisted in using high-water content cooking methods (e.g., stewing, steaming, boiling, poaching), instead of dry-heat methods (e.g., frying, grilling, roasting). In addition, the intervention group was provided with detailed written advice and counselling on how to choose foods low in AGEs and the amount and frequency of consumption allowed per day/week/month (e.g., choose a low-fat spread instead of butter - use 2 tsp 3-4/week). The goal was to reduce dietary AGE intake to <8000 kilounits (kU)/day.
Period: Overall Study
Arm/Group | Standard Diet - Control Group | Low AGE Diet - Intervention Group
Started | 19 | 19
Completed | 17 | 13
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Control group: Acute kidney injury requiring dialysis Intervention group: transplant rejection | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Diet - Control Group | Low AGE Diet - Intervention Group | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12) | 56 (10) | 56 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 12 | 15 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 16 | 16 | 32
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19 | 19 | 38
Skin autofluorescence [Mean (Standard Deviation); unit: Arbitrary units] — Tissue accumulation of advanced glycation end-products was assessed by measuring skin autofluorescence (SAF) using a validated Autofluorescence Reader. SAF is calculated as the ratio between emission and excitation and is expressed as arbitrary units (AU). Three measurements were conducted and the average value of these was used for statistical analysis. SAF reference value for the age group of 50-60 years is 2.1±0.4 AU
  Arbitrary units | 2.9 (0.6) | 3.0 (0.8) | 2.9 (0.7)
Dietary AGE intake [Median (Inter-Quartile Range); unit: Kilounits/day] | 17201 [13492 to 22551] | 20225 [16544 to 26004] | 18558 [15164 to 25341]

OUTCOME MEASURES:

1. Primary Outcome: Skin Autofluorescence (SAF) Levels at 6 Months
Description: Tissue accumulation of advanced glycation end-products was assessed by measuring skin autofluorescence (SAF) using a validated Autofluorescence Reader. SAF is calculated as the ratio between emission and excitation and is expressed as arbitrary units (AU). Three measurements were conducted and the average value of these was used for statistical analysis. SAF reference value for the age group of 50-60 years is 2.1±0.4 AU
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Standard Diet - Control Group | Low AGE Diet - Intervention Group
Number analyzed (Participants) | 17 | 13
Arbitrary units | 2.8 (0.6) | 2.8 (0.5)

2. Secondary Outcome: Participant Adherence to Diets
Description: Adherence to the low AGE diet (achieving dietary AGE intake <8000 kilounits [kU]/day) and the standard diet for persons with a kidney transplant was evaluated by means of a 3-day food diary (2 weekdays and 1 weekend day) every month (i.e., assessed from 1-6 months but only adherence at 6 months was reported).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Diet - Control Group | Low AGE Diet - Intervention Group
Number analyzed (Participants) | 17 | 13
Participants | 17 | 9

3. Secondary Outcome: Skin Autofluorescence (SAF) Trend.
Description: SAF was measured at baseline, 3 and 6 months. The rate of change of SAF among these 3 time points (i.e., SAF trend) was then calculated by fitting a regression line using the SLOPE function in Microsoft Excel 2016, where the y-axis represented SAF values and the x-axis represented time points.
Time Frame: 0, 3 and 6 months
Measure: Mean (Standard Deviation); unit: Arbitrary units/year
Arm/Group | Standard Diet - Control Group | Low AGE Diet - Intervention Group
Number analyzed (Participants) | 17 | 13
Arbitrary units/year | -0.22 (0.75) | -0.45 (1.19)

4. Secondary Outcome: Dietary AGE Intake at 6 Months
Description: A validated food frequency questionnaire was used to quantify the content of AGEs in foods.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: Kilounits/day
Arm/Group | Standard Diet - Control Group | Low AGE Diet - Intervention Group
Number analyzed (Participants) | 17 | 13
Kilounits/day | 20447 [14093 to 25044] | 5515 [4206 to 8631]

ADVERSE EVENTS:
Time Frame: 6 months.
Description: As a low-risk intervention, there was no requirement for non-serious adverse events (AEs) to be recorded or reported. However, any AEs that met the definition of serious (SAE) and are not listed below must be reported.
  Exceptions to SAE reporting:
  * Rejection
  * Infection
  * Graft Failure
  * New Onset Diabetes after Transplantation
  Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Standard Diet - Control Group | Low AGE Diet - Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT05104242/Prot_SAP_000.pdf